CLINICAL TRIAL: NCT02314533
Title: A Prospective, Open-label, Parallel, Controlled Study to Evaluate the Efficacy of Fenofibrate on Microalbuminuria in Hypertriglyceridemic Patients With Type 2 Diabetes on Top of Statin Therapy
Brief Title: Evaluate the Efficacy of Fenofibrate on Microalbuminuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, director of department of endocrinology, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FENOD003
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Microalbuminuria
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fenofibrate (Experimental): Fenofibrate 200mg capsule will be administered orally with breakfast once daily according to the Chinese prescription information of Lipanthyl, while previous type and dose of statin will be administered in the evening.
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate — Fenofibrate (Lipanthyl®) 200mg capsule will be administered orally with breakfast once daily
  Other Names: Lipanthyl

SUMMARY:
The investigators design this prospective, open-label, parallel, controlled study to investigate fenofibrate's effect on microalbuminuria reduction and serum creatinine on top of statin therapy in Chinese hypertriglyceridemic patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes has become a major public health problem in China, and a large-scale epidemiological survey revealed a prevalence of 9.7% approximately 5 years ago [1]. Diabetic nephropathy (DN) is the most common microvascular complication and is a major cause of end-stage renal disease that requires dialysis and/or renal transplantation [2]. Thus, strategies aimed at the treatment of DN are as important as those that target diabetes itself. Diabetic nephropathy is associated with mesangial cell expansion, thickening of glomerular and tubular basement membrane, glomerulosclerosis and tubular necrosis. These structural changes could lead to the occurrence of albuminuria, elevation of serum creatinine and urea nitrogen levels, and reduction in glomerular filtration rate[3].

Despite effective interventions such as angiotensin converting enzyme inhibitors and angiotensin-II-type 1(AT1) receptor blockers available to treat diabetic nephropathy[4-5], hitherto, no promising interventions are in the practice that could satisfactorily improve the clinical outcomes of diabetic nephropathy. Current treatment protocol for the management of diabetic nephropathy targets for tight glucose and blood pressure control as hyperglycemia and hypertension are major risk factors for the disease progression of nephropathy[6-7]. In addition, dyslipidemia has been suggested to be strongly associated with an induction and progression of diabetic nephropathy[8-9] While renal lipid accumulation- induced lipotoxicity could develop diabetic nephropathy[10], peroxisome proliferator-activated receptor a (PPARa) agonists could have a place in the treatment of diabetic nephropathy[11]. Experimental and clinical studies suggested that fenofibrate, a fibrate class of hypolipidemic agent, acts as a PPARa agonist, ameliorated diabetic renal damage by preventing renal oxidative stress, inflammation and fibrosis. Our previous studies showed that fenofibrate contributes its beneficial effect to prevent endothelial dysfunction from upregulating level of BH4 and decreasing production of ROS through the mechanism of increasing the level of intracellular GTPCH-I. Fenofibrate may help protect against vascular damage potential by promoting the re-coupling of eNOS with normalizing endothelial disorders[12-13]. Moreover, fenofibrate significantly reduced the pathological changes in glomeruli by improving the glomerular capillary size and reducing the mesangial expansion [14-16].

Few clinical studies have also confirmed the renoprotective potential of fenofibrate against diabetic nephropathy. The 'Fenofibrate Intervention for Event Lowering in Diabetes (FIELD)' study suggested that fenofibrate treatment had promising effects in preventing the progression of diabetes-associated microvascular complications, including diabetic nephropathy [17-18]. In the FIELD study, among all type 2 diabetic patients (9795 patients), over 5 years, the fell of ACR was greater in participants on fenofibrate (23.7% vs 11.5%), albuminuria on average progressed 14% less frequently and was reversed 18% more often among those diabetic patients received fenofibrate as compared to placebo.The investigators of this trial suggested that fenofibrate could protect against the loss of underlying renal function seen in patients with T2DM[19].And also in ACCORD study[20], a lower incidence of both micro- and macro-albuminuria was noted in the fenofibrate compared with the placebo group [38.2 vs. 41.6% (P = 0.01) and 10.5 vs. 12.3% (P = 0.04), respectively]. Unfortunately, during fenofibrate therapy in FIELD study, the plasma creatinine was noted to be increased, but quickly reversed on placebo assignment. Though it remained higher on fenofibrate treatment as compared to placebo, the chronic rise was slower with less loss of estimated glomerular filtration rate (eGFR). How these short-term increases can affect long-term renal function was also assessed in a retrospective subanalysis of the ACCORD study[21]. Among fenofibrate-treated patients, 321 experienced increased SCr levels>20% (cases) within the first 3 months of treatment. Patients with SCr increases <2% were controls (n = 175). In these patients as well as in 565 placebo-treated subjects, SCr and cystatin C levels were measured at baseline and 6-8 weeks after treatment discontinuation. As expected, cases had significantly higher SCr levels and lower eGFR than controls or placebo treated individuals at the end of the study. However, SCr levels and eGFR in cases returned to placebo levels 51 days after treatment discontinuation. At the same time, fenofibrate-treated patients with no initial increases in SCr levels had the lowest SCr levels and the highest eGFR. In the setting of careful renal function surveillance and reduction of fenofibrate dose as indicated, no increase in renal disease or cardiovascular outcome was seen in those individuals demonstrating fenofibrate-associated creatinine increase[22].Taken together, fenofibrate could delay albuminuria and eGFR impairment in T2DM patients. Of note, in a study reported by Hottelart et al. [23], fenofibrate associated increase in creatininemia in renal patients did not reflect an impairment of renal function. Fenofibrate-induced increase in creatinine production was suggested to be associated with an enhanced metabolic production rate of creatinine.

The Diabetes Atherosclerosis Intervention Study (DAIS) with patients of T2DM treated with micronized fenofibrate for an average of 38 months suggested that fenofibrate significantly reduced the worsening of albumin excretion, which was associated with reduced progression of normal albumin excretion to microalbuminuria [24]. The investigators concluded that the improvement in lipid profile with fenofibrate in patients with T2DM was associated with reduced progression to microalbuminuria.

These studies collectively suggest that fenofibrate could afford renoprotection and prevent the induction and progression of nephropathy in diabetic patients who are experiencing abnormal lipid profile and diabetic dyslipidemia with renal inflammation.

The investigators design this study to investigate fenofibrate's effect on microalbuminuria reduction and serum creatinine on top of statin therapy in Chinese hypertriglyceridemic patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Females or males, and aged 20 to 65 years.
* Type 2 diabetes with microalbuminuria (Urinary albumin /creatinine ratio, ACR, between 30 and 300 mg/g, a first morning spot urine sample will be used to approximate the 24-hour urine albumin excretion) in two consecutive laboratory tests before the study period.
* At least 2 months statin monotherapy with low to moderate dose (atorvastatin ≤20mg q.d. or rosuvastatin≤10mg q.d. or simvastatin≤40mg q.d. or pravastatin≤40mg q.d.or pitavastatin≤2mg q.d or fluvastatin≤80mg q.d.or lovastatin≤40mg q.d) prior to enrollemnt and plan to continue the same type and dose of statin.
* TG≥1.7 mmol/L (150mg/dl) and TG<5.65 mmol/L (500mg/dl).
* HbA1C<8% and blood pressure<140/90mmHg.

Exclusion Criteria:

* Any contraindication of fenofibrate and statins in Chinese label.
* Hepatic insufficiency (ALT or AST> 1.5*ULN)
* Renal insufficiency [Creatinine clearance rate (Ccr)]<60ml/min estimated from MDRD equation)
* CK > 1.5*ULN
* Hypothyroidism
* Use of non-statin lipid-regulating drugs such as niacin and fish oil in previous 1 month
* Combination use of other fibrates or drug with similar structure, especially ketoprofen
* Combination use of oral anticoagulants
* Pregnant or lactating woman
* Other conditions at investigator's discretion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
urinary albumin to creatinine ratio (mg/g) | 6 month

REFERENCES:
- [Derived] Sun X, Liu J, Wang G. Fenofibrate decreased microalbuminuria in the type 2 diabetes patients with hypertriglyceridemia. Lipids Health Dis. 2020 May 23;19(1):103. doi: 10.1186/s12944-020-01254-2. PMID 32446306